CLINICAL TRIAL: NCT06738784
Title: Evaluation of the Efficiency of the PRPP (Perceive, Recall, Plan and Perform) Task Analysis System on Support and Orientation Decisions for People With Aging Psychiatric Disorders (PATPV) Living in Independent Housing.
Acronym: ECO2PSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01961-46
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Mental Health; Aging Disorder; Psychiatric Disorder
Keywords: mental health; geriatric psychiatry; ergotherapy
MeSH Terms: conditions — Psychological Well-Being; Mental Disorders | interventions — Phosphoribosyl Pyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRPP Evaluation (Experimental): T0 to T3 months: Evaluations
  * Multi-professional assessment by mobile team or day hospital
  * Completion of PRPP on 2 activities
  T3 months: First referral
  - Decision on the participant's future orientation following the PRPP
  T3 months to T9 months: Outpatient psychosocial rehabilitation (standard care)
  * Personalized psychosocial rehabilitation program determined in part by the PRPP and carried out in the day hospital for all participants.
  * PRPP interventions (occupational therapy)
  T9 months: Reassessment and confirmation of orientation
  * Second round of PRPP based on activities assessed at T3 months
  * Questionnaires to help with referral decisions, completed by the multi-professional teams involved in the program, and by the treating psychiatrist after the second PRPP has been completed.
  Interventions: Behavioral: Perceive, Recall, Plan and Perform (PRPP) evaluation

INTERVENTIONS:
Behavioral: Perceive, Recall, Plan and Perform (PRPP) evaluation — Passing the PRPP for 2 activities

SUMMARY:
Over the past 30 years, mental health policy has been geared towards increasing the number of people receiving care in the community, with a reduction of over 50% in the number of general psychiatric beds. The WHO recommends the implementation of alternatives to hospitalization, through the development of outpatient and home-based psychiatric care programs that support independent living.

People suffering from psychiatric disorders show cognitive decline as they age, including deficits in perception, attention, memory and problem-solving. These cognitive problems affect the ability to carry out the tasks of daily life, and make it more difficult to remain at home. In order to avoid hospitalization for these psychiatrically-stabilized patients who are losing their autonomy, it is necessary to take into account their mental and cognitive handicap, and to provide them with appropriate compensation.

Occupational therapy is a discipline concerned with the assessment, rehabilitation and integration of people with disabilities. Occupational therapists provide ecological assessments to support personalized care plans. The PRPP (Perceive, Recall, Plan and Perform) task analysis system is a validated, ecological tool that integrates an occupational therapy assessment and intervention model. The PRPP assessment measures occupational performance and the impact of cognitive impairments on information processing and on the cognitive strategies required to carry out activities. Research conducted in Canada illustrates the value of PRPP in supporting people with schizophrenia. To the best of our knowledge, no team has studied the use of PRPP in the decision-making process for maintaining people with aging psychiatric disorders (PATPV) at home.

DETAILED DESCRIPTION:
The main hypothesis is that the use of the PRPP, through its scientific validity, will facilitate the decision-making of multi-professional care teams for the ambulatory support of PATPV to support :

* maintenance of independent housing
* or referral to a suitable place to live

This is a prospective, single-center study conducted within the "pathologies, handicap and aging" unit of the General and University Psychiatry (PGU) cluster at the Charles Perrens Hospital in Bordeaux.

The "pathologies, disability and aging" unit is dedicated to addressing the loss of autonomy and disability of people suffering from severe psychiatric disorders. One of its aims is to prevent hospitalization, particularly long-term hospitalization, for patients with chronic psychiatric pathologies who have become care-dependent. The program is structured around a multi-professional mobile team in charge of assessments, and a day hospital providing outpatient psychosocial rehabilitation care.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 40 years old
* Reside within the PGU sector (Mérignac, Pessac, Talence and Gradignan)
* Receive support from the PGU - CHCP "pathologies, disability and aging" department.
* Fluency in French

Exclusion Criteria:

* Being hospitalized for more than 18 months
* Refuse inclusion in the research project

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficiency of the PRPP system for living orientation | 9 months after inclusion
  Scoring the PRPP system for monitoring changes in occupational performance following the implementation of a personalized psycho-social rehabilitation project.

SECONDARY OUTCOMES:
Number of hospitalizations since inclusion | 12 months after inclusion
  Counting the number of hospitalizations

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Charles Perrens, Bourdeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chapparo, C., Ranka, J. L., & Nott, M. T. (2017). Perceive, Recall, Plan and Perform (PRPP) system of task analysis and intervention. In Occupational therapy for people experiencing illness, injury or impairment: Promoting occupation and participation (pp. 243-257). Elsevier
- [Background] Aubin G, Chapparo C, Gelinas I, Stip E, Rainville C. Use of the Perceive, Recall, Plan and Perform System of Task Analysis for persons with schizophrenia: a preliminary study. Aust Occup Ther J. 2009 Jun;56(3):189-99. doi: 10.1111/j.1440-1630.2007.00725.x. PMID 20854512
- [Background] Aubin G, Stip E, Gelinas I, Rainville C, Chapparo C. Daily activities, cognition and community functioning in persons with schizophrenia. Schizophr Res. 2009 Feb;107(2-3):313-8. doi: 10.1016/j.schres.2008.08.002. Epub 2008 Sep 27. PMID 18824328
- [Background] Lindstad MO, Obstfelder AU, Sveen U, Stigen L. Feasibility of the Perceive, Recall, Plan and Perform system of intervention for persons with brain injury in community-based rehabilitation: a pilot for a multiple-baseline design study. BMJ Open. 2023 Jun 28;13(6):e067593. doi: 10.1136/bmjopen-2022-067593. PMID 37380207
- [Background] Lindstad MO, Obstfelder AU, Sveen U, Stigen L. Effectiveness of the Perceive, Recall, Plan and Perform intervention for persons with brain injury in community-based rehabilitation: protocol for a single-case experimental design with multiple baselines. BMJ Open. 2022 Oct 5;12(10):e060206. doi: 10.1136/bmjopen-2021-060206. PMID 36198473